CLINICAL TRIAL: NCT04362891
Title: Safety, Longevity and Patient Satisfaction Comparison of Four Hyaluronic Acid Soft Tissue Fillers in Lip Augmentation: Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Four Hyaluronic Acid Fillers for Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Faceland Clinics (Other)
Responsible Party: Principal Investigator, Prof. dr. J. de Lange, Prof. dr. J. de Lange, Head of OMFS Surgery, Principal Investigator, Clinical Professor, at AUMC - location AMC, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL73349.029.20
Record Dates: First submitted 2020-04-16; First posted 2020-04-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Lip
Keywords: Hyaluronic Acid; Dermal Fillers; Lip; Safety; Longevity; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Multicenter; triple blind; randomized; parallel; controlled trial with 4 treatment arms (4 different widely used commercially available HA soft tissue fillers with FDA approval status and/or CE-marking for cosmetic facial use).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcome Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Juvéderm® (Experimental): Cross-linked hyaluronic acid dermal filler product brand A (1,0 mL at baseline and 0,2 mL touch-up at 2-week follow-up).
  Interventions: Procedure: Cosmetic lip augmentation
- Restylane® (Experimental): Cross-linked hyaluronic acid dermal filler product brand B (1,0 mL at baseline and 0,2 mL touch-up at 2-week follow-up).
  Interventions: Procedure: Cosmetic lip augmentation
- Belotero® (Experimental): Cross-linked hyaluronic acid dermal filler product brand C (1,0 mL at baseline and 0,2 mL touch-up at 2-week follow-up).
  Interventions: Procedure: Cosmetic lip augmentation
- Stylage® (Experimental): Cross-linked hyaluronic acid dermal filler product brand D (1,0 mL at baseline and 0,2 mL touch-up at 2-week follow-up).
  Interventions: Procedure: Cosmetic lip augmentation

INTERVENTIONS:
Procedure: Cosmetic lip augmentation — The primary study treatment site will be the vermilion (body of the lip); additional areas (vermilion borders, Cupid's bow, philtral columns, and/or oral commissures) will be treated if deemed appropriate by the treating physician. Treatment will be administered through intradermal, subdermal, and/or intramuscular injection within the orbicularis oris muscle. Injection techniques for each area will include linear threading, serial puncture, fanning, and/or cross-hatching. The treating physician will determine the appropriate volume to inject based on clinical experience and the subject's goals for lip augmentation.

SUMMARY:
There is need for evidence-based and reproducible data comparing the safety, longevity and patient satisfaction propensity of the various HA soft tissue filler products. Among cosmetic HA soft tissue filler procedures, especially the lip augmentation has become common. Therefore, the aim of this study is to determine whether a statistically significant difference can be detected in the safety, longevity and/or patient satisfaction related to four HA soft tissue filler products widely used for cosmetic lip augmentation. Specifically, the aim of this study is to determine whether superiority of one or more product(s) over the others can be detected.

DETAILED DESCRIPTION:
Rationale: Currently, hyaluronic acid (HA) soft tissue fillers are widely employed in cosmetic medical practice for facial contouring and rejuvenation. Among these procedures, especially the lip augmentation has become common. To this end various products have become commercially available, however to date no robust evidence is available to support the safety, longevity or patient satisfaction propensity superiority of one product over the others.

Objective: To assess whether superiority in safety, longevity and patient satisfaction propensity can be shown of one of four most frequently used FDA-approved and/or CE marked HA fillers worldwide, used to augment the lip, over the others.

Study design: Multi-center, randomized, controlled, four group, parallel, triple-blind clinical trial of 160 adult participants.

Study population: Consecutive healthy individuals with no history of previous lip treatment and a self-reported wish for lip augmentation, who present at one of the private cosmetic medicine clinics in the Netherlands, will be recruited.

Intervention (if applicable): After giving informed consent, participants will be randomized to receive a protocoled lip augmentation procedure by the injection of either 1 mL of brand A, B, C or D.

Main study parameters/endpoints: The primary outcome measure will be the absolute lip volume augmentation as measured by the Lemperle Lip Index from baseline to 3-months follow-up. Secondary outcomes will include the incidence of serious adverse reactions and side effects related to the procedure, the absolute volume augmentation from baseline to 2-weeks follow-up and self-reported quality of life and satisfaction with aesthetic results from baseline to 2-weeks follow-up as measured by validated FACE-Q questionnaire scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over.
* Female sex.
* No history of previous lip augmentation treatment.
* Oral and written informed consent to participate in the study.
* Desire for cosmetic lip augmentation to improve one's physical or mental well-being.
* Actively treatment seeking (patient actively chooses to make an appointment at a Faceland private cosmetic clinic without invitation).
* Small to moderately full lip volume (Merz Lip Scale score 0 - 2 out of 4).

Exclusion Criteria:

* Active peri-oral infection in vicinity of injection site
* Tumour in vicinity of injection site
* Active tuberculosis
* Pregnant or breast-feeding
* History of severe hypersensitivity to filler components (sodium hyaluronate preparations or local anesthetics of the -amide type, gram-positive proteins, wasps/bees or the hyaluronidase enzyme)
* Active collagenosis (e.g., active systemic lupus)
* Graft vs. host disease
* Active Hashimoto's disease
* Use of thrombolytics or anticoagulants with high bleeding risk
* General infection
* Porphyria
* Untreated epilepsy
* Keloid tendency
* Cardiac arrythmia
* Severe liver or kidney disease
* Fulfilling the DSM-5 diagnostic criteria for Body Dyspmorphic Disorder
* Concurrent laser- peeling- or dermabrasia treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Longevity of absolute lip volume augmentation | from baseline to 3-months follow-up
  The primary outcome will be the longevity of the absolute lip volume augmentation, as measured by the modified Lemperle Lip Index (vertical height in mm).

SECONDARY OUTCOMES:
Patient satisfaction (lip appraisal) | from baseline to 3-months follow-up
  Patient satisfaction with the treatment as measured by validated FACE-Q questionnaire "Lips" score.
Quality of Life (Social) | baseline to 3-months follow-up
  Quality of Life as measured by validated FACE-Q questionnaire "Social Function" score.
Quality of Life (Psychological) | baseline to 3-months follow-up
  Quality of Life as measured by validated FACE-Q questionnaire "Psychological Wellbeing" score.
Product safety (serious adverse events) | baseline, 2-weeks and 3-months follow-up
  Product safety, as measured by serious adverse events related to the procedure.

OTHER OUTCOMES:
Effectiveness of absolute lip volume augmentation at week 2 | from baseline to 2-weeks follow-up
  A between-group difference in volume augmentation from baseline to 2-weeks follow-up,
Patient satisfaction (with treatment outcome) | at 2 weeks and 3 months follow-up
  Patient satisfaction with the treatment as measured by validated FACE-Q questionnaire scores "Satisfaction with Outcome of Treatment" score.
Patient satisfaction (with decision) | at 2 weeks and 3 months follow-up
  Patient satisfaction with the treatment as measured by validated FACE-Q questionnaire "Satisfaction with Decision to Have Treatment" score.
Side-effects (psychological impact of recovery from treatment) | at 2 weeks and 3 months follow-up
  Side-effects, as measured by the FACE-Q questionnaire "Early Life Impact" score.
Side-effects (physical discomfort) | baseline, 2-weeks and 3-months follow-up
  Side-effects, as measured by the FACE-Q questionnaire "Adverse Effects Lips" score.
Side-effects (recovery of side-effects) | baseline, 2-weeks and 3-months follow-up
  Side-effects, as measured by validated FACE-Q questionnaire scores "Recovery Early Symptoms" score.
Absolute lip volume augmentation at week 2 | from baseline to 2-weeks follow-up
  The absolute lip volume augmentation as measured by the Lemperle Lip Index.

CONTACTS AND LOCATIONS:
Overall Officials: Jan de Lange, MD DDS PhD, Principal Investigator — University of Amsterdam
Locations (4):
- Netherlands (4):
  - Faceland Almere, Almere Stad, Flevoland
  - Faceland Eindhoven, Eindhoven, North Brabant
  - Faceland Rotterdam, Rotterdam, South Holland
  - Faceland Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stojanovic L, Majdic N. Effectiveness and safety of hyaluronic acid fillers used to enhance overall lip fullness: A systematic review of clinical studies. J Cosmet Dermatol. 2019 Apr;18(2):436-443. doi: 10.1111/jocd.12861. Epub 2019 Jan 12. PMID 30636365
- [Result] Alam M, Kakar R, Nodzenski M, Ibrahim O, Disphanurat W, Bolotin D, Borovicka JH, Pace N, Alster TS, Arndt KA, Beer KR, Berlin JM, Bernstein LJ, Brightman LA, Butterwick K, Cox SE, Chotzen V, Fabi SG, Fitzpatrick RE, Geronemus RG, Goldman MP, Groff WF, Kaminer MS, Kilmer S, Rohrer TE, Tanzi EL, Silva SK, Yoo SS, Weinkle SH, Strasswimmer J, Poon E, Dover JS. Multicenter prospective cohort study of the incidence of adverse events associated with cosmetic dermatologic procedures: lasers, energy devices, and injectable neurotoxins and fillers. JAMA Dermatol. 2015 Mar;151(3):271-7. doi: 10.1001/jamadermatol.2014.2494. PMID 25372511
- [Result] Barone M, Cogliandro A, Cagli B, Persichetti P. FACE-Q Scales for Health-Related Quality of Life, Early Life Impact, Satisfaction with Outcomes, and Decision to Have Treatment: Development and Validation. Plast Reconstr Surg. 2015 Aug;136(2):272e-273e. doi: 10.1097/PRS.0000000000001439. No abstract available. PMID 26218401